CLINICAL TRIAL: NCT02705833
Title: Head and Neck Cancer Treatment Patterns and Outcomes Research Study in France, Germany, and Canada
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-551
Record Dates: First submitted 2016-02-25; First posted 2016-03-11 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Population with R/M SCCHN: Recurrent/Metastatic (R/M) Squamous Cell Carcinoma of the Head and Neck (SCCHN) patients diagnosed between 01July2013 and 30June2014, alive or deceased, at the time of data collection

SUMMARY:
The primary objective of the study is to characterize the medical management of squamous cell carcinoma head and neck (SCCHN) patients diagnosed with recurrent/metastatic (R/M) disease (between 01July2013 and 30 June 2014) in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years old or older) with a confirmed diagnosis or R/M head and neck, may be living or deceased at time of enrollment in the study
* Diagnosis of R/M head and neck cancer between 01July2013 and 30June2014 (study index period)

Exclusion Criteria:

* If female patient, pregnant or lactating between 01July2013 and 30June2014
* Enrolled in cancer treatment-clinical trials since diagnosis of R/M head and neck cancer during the study index period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with R/M SCCHN between 01July2013 and 30June2014
Sampling Method: Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Best Therapy Response defined as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD) based on physician's assessment for each therapy regimen | approximately 12 months
Overall Survival(OS) of patients with an Index diagnosis of R/M SCCHN | approximately 12 months
Progression-Free Survival(PFS) of patients with an Index diagnosis of R/M SCCHN | approximately 12 months
Recurrent-Free Survival(RFS) of patients with an Index diagnosis of R/M SCCHN | approximately 12 months
Overall Response Rate(ORR) of patients with an Index diagnosis of R/M SCCHN | approximately 12 months

SECONDARY OUTCOMES:
Frequency of R/M SCCHN-related health care resource use | approximately 12 months
Treatment selection conditional on patient demographics, comorbidities, disease severity, and other characteristics as well as clinician demographics, therapy preferences, and other characteristics | approximately 12 months
Best Therapy Response conditional on patient demographics, comorbidities, disease severity, treatment received, and other characteristics | approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx